CLINICAL TRIAL: NCT01575249
Title: Prospective Study Focused on idEntification of cliNical, Biological and Imagistic Parameters in rapId-proGression Subgroup Patients With Moderate Aortic Stenosis
Brief Title: Identification of Parameters in rapId-proGression Subgroup Patients With Moderate Aortic Stenosis
Acronym: ENIGMAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, MISCHIE Nicolae Alexandru, CARDIOLOGIST, ASSISTANT PROFESSOR, Carol Davila University of Medicine and Pharmacy
Other Study IDs: The ENIGMAS trial
Record Dates: First submitted 2012-04-09; First posted 2012-04-11 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Aortic Stenosis
Keywords: progression; moderate aortic stenosis; asymptomatic; symptomatic
MeSH Terms: conditions — Aortic Valve Stenosis; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — standard blood count, c-reactive protein, urea, creatinin, hepatic standard biology, serum calcium, cholesterol and tryglicerides.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asymptomatic group: one hundred patients with a negative exercise stress echo for symptoms/ECG/wall motion abnormalities (WMA), negative spirometry test for pulmonary disease, without known CAD or other valvular diseases, in sinus rhythm and with a LVEF>55%
- Symptomatic group: one hundred patients with symptomatic AS (negative pulmonary tests but positive stress echo or prior CAD or other valvular diseases and a LVEF>55%

SUMMARY:
The investigators aim to identify all clinical, biological, echo and imagistic parameters that predispose to increased progression rates in a prospective observational trial which will include ONLY patients with moderate AS, with the complete cardiological investigational tools provided in 2012. Once those parameters are found, medical and interventional treatment could be implemented to decrease the mortality rates.

DETAILED DESCRIPTION:
1. Why this study? 1.1. Significance and difficulty of the problem being addressed. Aortic stenosis is the most encountered valvular disease According to the 2007 ESC guidelines (1), moderate aortic stenosis (AS) is defined as valve area 1.0-1.5 cm² (0.6 cm²/m² to 0.9 cm²/m² body surface area (BSA)) or mean aortic gradient of 30-50 mmHg in the presence of normal flow conditions. We already know how to treat patients with severe AS, symptomatic or not. On the contrary, in patients with moderate AS there is not a clear agreement on what to do to reduce the excess mortality (detailed below). Why do these patients die and what can we do to reduce mortality rates? 1.2. Originality of the proposed solution and the appropriateness of the objectives. There are already some progression factors in all spectrum of AS that have been highlighted (discussed below) and which could influence mortality in this patient subgroup, but none of the studies address exclusively to moderate AS. The majority of these studies have major limitations, are not prospective, and even if some are, the parameters followed do not cover the complete cardiological investigational tools (no 3D left ventricular (LV) ejection fraction (EF), no strain, no magnetic resonance imaging (MRI), etc.). As in any major disease, lots of studies that include moderate AS are contradictory on the same matter (see progression of AS). We aim to identify all clinical, biological, echo and imagistic parameters that predispose to increased progression rates in a prospective randomized trial which will include ONLY patients with moderate AS, with the investigational tools provided in 2012. Once those parameters are found, medical and interventional treatment could be implemented to decrease the mortality rates.

   But first, some data about survival and death in moderate AS. I would like to start by paraphrasing one of the most passionate researchers in the field of aortic stenosis, C. Otto (2): "even mild disease is important" (referring of course at the outcomes of patients with mild AS). Similarly, people with moderate AS/ aortic sclerosis, not even mentioning moderate to severe AS (3) have an increased death rate in comparison to age-matched healthy population. The same author reported in 1999 the results of a prospective study (4) with a follow-up (FU) at 5 years and she observed a cardiac death rate of 6.1% in general population (normal aortic valves), 10.1% in patients with aortic sclerosis and 19.6% in patients with AS. In 2004 Rosenhek et al. (5) found a cardiac death rate of 8.7% in a population with mean age of 67 years, with moderate AS at the initial examination. Even though the largest study (6) evaluating medical treatment in moderate AS reported a cardiac death rate of 6.0% (similar to general population), we consider this study not eloquent because there was a super-selected population enrolled (investigators ruled out the most important progression factors of AS: exclusion criteria included history of coronary artery disease (CAD), stroke and diabetes mellitus (DM)).
2. Trials involving patients with moderate AS. In this presentation we will not review or discuss outcomes of severe AS, but ONLY outcomes of patients with MODERATE AS.

   The first step in our research was the identification of all studies involving moderate AS. We observed that there are few studies that included ONLY patients with moderate AS. At the opposite, the large majority of studies included moderate AS among all spectrum of AS patients (sclerosis, mild, moderate, severe- alone or combined). That is why we categorized all previous studies regarding moderate AS by the baseline inclusion criteria. We found 4 major groups of enrolled patients that we reviewed and discussed below: patients with mild to moderate AS (Table 1) (5-10), patients with moderate AS (Table 2)(11-12), patients with mild, moderate and severe AS (Table 3)(13-20) and patients with moderate to severe AS (Table 4)(21-27).

   Even though all essential data regarding moderate AS can be easily read in the tables (patient characteristics, progression of moderate AS, outcomes, survival, limitations and conclusions) and even though progression factors are summed-up below, of great importance are the results of some echo studies recently published on which I would like to briefly discuss. Monin et al. enrolled 107 patients with baseline peak velocity (PV) of 3.5 to 4.4 m/s (26), he concluded that female sex, PV and brain natriuretic peptide (BNP) at baseline were correlated with AS progression and developed a score to best stratify outcomes in these patients (see Table 4 for limitations). Marechaux et al. (27) included 135 patients with at least moderate AS (53% had severe AS), with normal stress test at baseline. Increased progression was present in those with resting mean gradient (MG) >35 mmHg and exercise-induced increase in MG >20 mmHg (see Table 4 for limitations). Two studies tried to clarify the role of strain in AS. One of the studies showed that strain gradually decreased as severity of AS increases and that global longitudinal strain (GLS) might be useful to assess subtle changes in LV function in patients with mild, moderate and severe AS (17). In the second study, Ng et al. (19) found that longitudinal, radial and circumferential strain and strain rate (SR) deteriorate with aortic valve disease progression. Important limitations of both studies are found in Table 3.
3. Progression of AS. There is a wide variability in AS progression. Progression rates (for the PV) begin from 0.15±0.01 m/s/y in population without cardiovascular risk factors (6) and increase to 0.34±0.42 m/s/y in patients with CAD, reaching 0.45±0.38 m/s/y in patients with cardiovascular events (5).

   High progressors are those that have at least one abnormal parameter of the followings: echocardiography parameters: baseline PV (3, 12, 5, 10, 16, 20, 26), baseline peak gradient (24), mean gradient (3), rate of increase in PV (3, 20), moderate to severe aortic valve calcification on echo (5, 12), LV hypertrophy (27), resting MG >35 mmHg (27), exercise-induced increase in MG >20 mmHg (27), E velocity (16), bicuspid aortic valve (16); clinical predictors: CAD (5, 21), age (>80 years-8, 12, 18, 20, >64 years-21, >65years-27), diabetes (14, 27), metabolic syndrome (MS) (24), dialysis (28, 29), increased BMI (7), functional status (3), history of smoking (7, 30), systolic blood pressure (SBP) (18, 30), male gender (24, 30), female gender (26); and biological parameters: parathyroid hormone (PTH) level (18), BNP at baseline (26), high lipoprotein (a) (Lp(a)) and low density lipoprotein (LDL) cholesterol levels (30).

   No influence on AS progression were treatment with simvastatin and ezetimibe (6), elprenone (25) or rosuvastatin (9) and statins (14).

   Slower progression was observed after osteoporosis (11) and bisphosphonate treatment (15), but studies were either too small, retrospective (11, 15) or biased (11). Geographical differences are evident in two papers which show that Korean patients progress slower than western population (12, 16).

   Data regarding the role of C-reactive protein in AS progression are controversial (10, 13).

   We did not discuss the old studies or small series of patients with AS, some in the era of cardiac catheterizations (31-36), some in the early echo decades (37-41). Their capability to address this subject was limited by a retrospective design in most cases, potential selection bias, limited clinical, functional, or exercise data, the availability of only two data points per patient, lack of factors that predict the rate of hemodynamic progression and clinical outcome.
4. Incidence of AS. Degenerative aortic valve disease evolves slowly from aortic sclerosis to aortic stenosis. Aortic sclerosis and stenosis are found in about 29% and 2-9% respectively in adults older than 65 years (4). In 5,201 subjects > 65 years, aortic valve sclerosis was present in 26% and AS in 2% of the entire study cohort; in subjects >75 years of age, sclerosis was present in 37% and stenosis in 2.6% (30). The prevalence of critical AS was 2.9% in the group 75 to 86 years of age in another study (42). In an observational study (43) which enrolled 953 subjects (aged 25-74 years), the overall prevalence of degenerative aortic valve disease (defined as the presence of valvular sclerosis, calcification, or thickening on echocardiographical examination) was 28%. The prevalence of degenerative aortic valve disease by age groups was the following: 7% (35-44 years), 19% (45-54), 30% (55-64), 38% (65-74) and 64% (75-84). There were no significant differences between men and women.

Clinical factors associated with AS are similar to those associated with CAD (3, 44). Even though several small non-randomized studies (45, 46-49) suggested a beneficial effect of statins, three prospective randomized studies did not find any effect of lipid-lowering therapy on the progression of aortic-valve stenosis.(6, 10, 50).

ELIGIBILITY:
Inclusion Criteria:

* age 21 years;
* native aortic valve leaflet thickening with reduced systolic opening on two-dimensional echocardiography and an aortic jet velocity at rest between 2.8 and 3.1 m/s or a valve area calculated by the continuity equation of 1.7 to 1.5 cm2, evaluated at a heart rate between 60 and 90/ minute and at a systolic arterial pressure of 120-140mmHg at baseline;
* LVEF > 55% (calculated by modified Simpson formula).

Exclusion Criteria:

* positive stress test (symptoms including dyspnoea, angina, syncope, ECG pathological changes, WMA);
* positive pulmonary disease (spirometry);
* heart failure;
* LVEF < 55%;
* moderate/severe aortic or mitral regurgitation or mitral stenosis, subvalvular or supravalvular AS, dynamic subaortic obstruction;
* CAD (history of MI or coronary artery stenosis on coronary angiography);
* active endocarditis;
* rhythm other than sinus rhythm;
* severe uncontrolled risk factors for CAD:

  * uncontrolled DM,
  * uncontrolled hypertension (SBP > 180mmHg),
  * refuse to discontinue smoking,
  * persistent hypercholesterolemia under treatment (total cholesterol > 240mg/dl);
* glomerular filtration rate < 30% or patient requiring dialysis;
* patient refusal; survival expectancy < 2 years;
* inability to perform physical exercise;
* suboptimal echo window;
* different types of echo machines.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrollment will be done by echo screening of the population (of the 3rd Arrondissement in Bucharest, Romania) with age >50 years until target patients reached and also by screening out-patients arriving at "Bagdasar-Arseni" Emergency Hospital (Bucharest) with other cardiovascular diseases other than specified in the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
occurrence of major adverse cardiac events (MACE) defined by the followings: death, aortic valve replacement (AVR) and myocardial infarction (MI). | 3 years

SECONDARY OUTCOMES:
TIME TO SYMPTOMS (angina, dyspnea, syncope) at stress echocardiography | 3 years
TIME TO ALTERED HEMODYNAMIC PARAMETERS at stress (strain decrease, EF decrease, ventricular arrhythmia, decrease in SBP, stress gradients suggestive of severe AS) | 3 years
differentiate outcomes of patients with mean gradients between 40 and 50 mmHg (grey zone of AS) | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDRU N MISCHIE, MD, Principal Investigator — BAGDASAR ARSENI EMERGENCY HOSPITAL
Locations (1):
- "Bagdasar-Arseni" Emergency Hospital, Bucharest, Romania

REFERENCES:
- See also: protocol of the SEAS trial — http://www.ncbi.nlm.nih.gov/pubmed?term=6.%20Rosseb%C3%B8%20AB%2C%20Pedersen%20TR%2C%20Boman%20K%2C%20Brudi%20P%2C%20Chambers%20JB%2C%20Egstrup%20K%2C%20Gerdts%20E%2C%20Gohlke-B%C3%A4rwolf%20C%2C%20Holme%20I%2C%20Kes%C3%A4niemi%20YA%2C%20Malbecq%20
- See also: similar protocole to our study — http://www.ncbi.nlm.nih.gov/pubmed?term=Usefulness%20of%20exercise-stress%20echocardiography%20for%20risk%20stratification%20of%20true%20asymptomatic%20patients%20with%20aortic%20valve%20stenosis.